CLINICAL TRIAL: NCT02924935
Title: Histidine Therapy: A Project to Treat HARS Deficiency
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108364
Record Dates: First submitted 2016-09-16; First posted 2016-10-05 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: HARS Syndrome
MeSH Terms: interventions — Histidine

STUDY DESIGN:
Intervention Model Description: Participants are given L-Histidine supplements and were prescribed to take 50mg/kg twice daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): L-Histidine in 500mg capsules taken at a dose of 50mg/kg to maintain high-normal serum histidine levels
  Interventions: Dietary Supplement: L-Histidine

INTERVENTIONS:
Dietary Supplement: L-Histidine — L-Histidine in 500mg capsules taken at a dose of 50mg/kg to maintain high-normal serum histidine levels

SUMMARY:
This study evaluates the role of histidine in patients with HARS Syndrome. Children with HARS Syndrome will receive oral nutritional supplementation with histidine at a dose which will be increased in the event of acute febrile illness. Vision, hearing and plasma biomarkers will be monitored throughout the study period.

DETAILED DESCRIPTION:
HARS syndrome is a progressive degenerative disease affecting eyesight and hearing caused by a mutation in the HARS gene which codes for an enzyme involved in protein synthesis. HARS syndrome has been exclusively found in the Old Order Amish communities in Southwestern Ontario and in Pennsylvania. Children with this disorder initially have normal vision and hearing, but with a febrile illness, can have a sudden loss of vision and hearing, as well as visual hallucinations. There is some evidence that vision loss progresses, albeit at a slower rate, even without a febrile incident. In more severe cases, fluid accumulates in the lungs (acute respiratory distress syndrome or ARDS) which can cause a drop in oxygen levels and sometimes death. There is currently no specific treatment for HARS syndrome, apart from supportive care. Anecdotal evidence of an adult with HARS syndrome who was treated with the amino acid L-histidine suggests that there was an improvement in vision, however there were no baseline objective measurements of vision prior to the use of histidine. We have designed a pilot project in which histidine will be given to children with HARS for 6 months. Investigators hypothesize that the histidine will be well tolerated and easily administered, without side effects. Investigators will monitor vision, hearing and bloodwork to determine if there is any change during the course of treatment. As well, investigators plan to administer increased doses of histidine during acute illnesses, hoping to prevent deterioration in breathing due to ARDS. The results of this initial pilot project may pave the way for a longer term study of the use of histidine.

ELIGIBILITY:
Inclusion Criteria:

1. Have molecularly confirmed HARS syndrome (Y454S homozygous).
2. Capable of giving informed consent or assent, or have an acceptable surrogate capable of giving consent on the participant's behalf.
3. Participant or surrogate decision maker is able to understand the study procedures and comply with them throughout the course of the study.
4. Able to take solid foods (ie applesauce) or swallow capsules (in younger children, capsule may be broken and contents mixed with applesauce).
5. At least 1 year of age or greater than 8 kg in weight (since histidine is supplied as a minimal dose of 500 mg/capsule.

Exclusion Criteria:

1. Unable or unwilling to give informed consent.
2. Unable to understand instructions or unable to attend clinic visits.
3. Children less than 1 year of age or less than ~8kg in weight (since histidine is supplied as 500 mg capsules).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity maintenance or improvement | 2 years
  Changes from baseline eye exam
Visual acuity maintenance or improvement | 2 years
  Changes from baseline electroretinography
Visual acuity maintenance or improvement | 2 years
  Changes from baseline ocular coherence tomography
Auditory ability maintenance or improvement | 2 years
  Changes from baseline auditory brainstem response
Auditory ability maintenance or improvement | 2 years
  Changes from baseline autoacoustic emissions
Auditory ability maintenance or improvement | 2 years
  Changes from baseline routine ear exam
Auditory ability maintenance or improvement | 2 years
  Changes from baseline audiometry
Changes in severity of acute febrile illness | 2 years
  Measured by length of hospital stay
Changes in severity of acute febrile illness | 2 years
  Measured by requirement for intensive care unit transfer
Changes in severity of acute febrile illness | 2 years
  Measured by number of hospitalizations

SECONDARY OUTCOMES:
Biomarker Changes | 2 years
  Changes to inflammatory markers, HARS protein, HARS antibodies, Amino acid levels and biochemical markers as a result of histidine therapy
Plasma level maintenance | 1 month
  Does histidine supplementation result in increased plasma histidine levels

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, Department of Paediatrics, Division of Medical Genetics, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No